CLINICAL TRIAL: NCT01243008
Title: A Single Centre, Randomized, Investigator Blinded, Placebo-controlled Ascending Dose Study to Assess the Local Safety, the Skin and Plasma Concentration of Azithromycin Dermal Formulation During Repeated Applications on the Skin of Healthy Volunteers
Brief Title: Safety, Skin and Plasma Concentration of Azithromycin Dermal Formulation
Acronym: IXO-01
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Ixodes GmbH (Unknown); Appletree AG (Industry)
Responsible Party: Thomas Kündig, University Hospital Zurich
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: IXO-01
Record Dates: First submitted 2010-09-16; First posted 2010-11-17 (Estimated); Last update posted 2010-11-19 (Estimated); Status verified 2010-11

CONDITIONS: Lyme Disease
Keywords: Lyme disease; Borreliosis; Azithromycin
MeSH Terms: conditions — Lyme Disease; Borrelia Infections

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Application of SHB001 — * Cohort 1: Application of SHB001 on the skin of right thigh
  * Cohort 2:
    1. Application of SHB001 on the skin of right thigh
    2. punch biopsies of treated skin areas
  Other Names: 0% SHB001 azitrhomycin dermal formulation (placebo); 5% SHB001 azitrhomycin dermal formulation; 10% SHB001 azitrhomycin dermal formulation

SUMMARY:
IXODES GmbH intends to develop SHB001, an azithromycin dermal formulation in order to prevent Lyme disease at early stages of infection after tick bite.

DETAILED DESCRIPTION:
In this study two consecutive cohorts will be treated:

* Cohort 1: 8 volunteers
* Cohort 2: 24 volunteers, divided into 3 groups of 8 subjects each

The study will be conducted in the following three phases:

1. Treatment of cohort 1: The aim is to establish the maximal tolerated dose (MTD) for a local treatment with azithromycin dermal formulation.

   1. Treatment of cohort 1 with azithromycin dermal formulation and follow up
   2. Assessment of local safety within the 7 days following the first treatment
   3. The maximal tolerated dose (MTD) will be determined
2. Treatment of cohort 2: The aim is to confirm the local tolerance of the selected doses and to evaluate the local skin and plasma concentration of azithromycin after application of SHB001 dermal formulation.

   1. Treatment of cohort 2 with azithromycin dermal formulation at maximal tolerated dose (MTD), with a dose one or more concentrations lower than maximal tolerated dose (MTD) and with placebo
   2. Skin biopsies of treated skin areas will be taken for the PK assessment
3. Study completion examination

ELIGIBILITY:
Main inclusion criteria:

* Male or female healthy volunteers, age 18 - 70 years

Main exclusion criteria:

* A known hypersensitivity against azithromycin, erythromycin or any of the macrolide antibiotics
* A known hypersensitivity against lidocaine
* Treatment by any route with any macrolide antibiotic within the last 2 month

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-04; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Local safety | April 2010 - November 2010
  The primary objective of this study is to assess the local safety of azithromycin dermal formulation when applied to healthy skin in healthy volunteers. This will be done by determination (in cohort 1) and confirmation (in cohort 2) of the maximal tolerated dose (MTD) after dermal application of SHB001 in 4 different dose regimens.

SECONDARY OUTCOMES:
Pharmacokinetics of SHB001 | April 2010 - November 2010
  * To assess the pharmacokinetics of azithromycin dermal formulation in the plasma in healthy volunteers after daily administration for three consecutive days in cohort 1 and cohort 2.
  * To assess the pharmacokinetics of azithromycin dermal formulation in the skin in healthy volunteers after daily administration for 1 - 3 consecutive days in cohort 2 only.
  * To demonstrate that the Minimal Inhibitory Concentration (MIC) of B.b. (=0.03μg/ml) in the skin is reached at least for 2 consecutive assessments (biopsies) in cohort 2.
  * To assess general safety in cohort 1 and 2.

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich
Locations (1):
- Clinical Trials Center, University and University Hospital Zurich, Zurich, Canton of Zurich, Switzerland